CLINICAL TRIAL: NCT07309952
Title: Neoadjuvant Stereotactic Body Radiotherapy Followed by Sintilimab Plus Chemotherapy for Locally Advanced Non-Small Cell Lung Cancer With Contralateral Mediastinal (N3) Lymph Node Metastasis: A Prospective Phase II Clinical Trial
Brief Title: Neoadjuvant SBRT Followed by Sintilimab Plus Chemotherapy for N3-Positive NSCLC
Acronym: SACTION 2501
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yang Hong (Other)
Responsible Party: Sponsor-Investigator, Yang Hong, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2025-696-01
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Locally Advanced Non-Small Cell Lung Cancer; Stage IIIb Non-small Cell Lung Cancer; Stage IIIC Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sintilimab; Paclitaxel; Carboplatin; Pemetrexed; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental : neoadjuvant SBRT combined with immunochemotherapy (Experimental)
  Interventions: Drug: Sintilimab; Drug: Paclitaxel; Drug: Carboplatin (AUC 5); Drug: Pemetrexed 500 mg/m2; Radiation: Stereotactic body radiotherapy (SBRT); Procedure: non-small cell lung cancer

INTERVENTIONS:
Drug: Sintilimab — Sintilimab is an anti-PD-1 monoclonal antibody. In this study, it is administered intravenously at a fixed dose of 200 mg on Day 1 of each 3-week cycle. Patients receive 2 cycles of sintilimab in combination with platinum-based doublet chemotherapy. The first dose of sintilimab is initiated within 7 days after completion of stereotactic body radiotherapy (SBRT).
Drug: Paclitaxel — Paclitaxel is a taxane chemotherapeutic agent. In this study, it is specifically used for patients with squamous cell non-small cell lung cancer (NSCLC). It is administered intravenously at a dose of 175 mg/m² on Day 1 of each 3-week cycle. Patients receive 2 cycles of paclitaxel in combination with sintilimab (anti-PD-1 antibody) and carboplatin (platinum-based agent) as part of the neoadjuvant regimen. Standard premedication to prevent hypersensitivity reactions is required prior to each infusion. This systemic chemotherapy phase is initiated within 7 days after the completion of stereotactic body radiotherapy (SBRT) to the primary lung tumor.
Drug: Carboplatin (AUC 5) — Carboplatin is a platinum-based chemotherapeutic agent. In this study, it serves as the backbone chemotherapy for all patients, regardless of histology. It is administered intravenously on Day 1 of each 3-week cycle. The dose is calculated using the Calvert formula to achieve a target area under the concentration-time curve (AUC) of 5 mg/mL/min. Patients receive 2 cycles of carboplatin in combination with sintilimab (anti-PD-1 antibody) and either pemetrexed (for non-squamous NSCLC) or paclitaxel (for squamous NSCLC). This chemoinmunotherapy phase commences within 7 days after the completion of stereotactic body radiotherapy (SBRT) to the primary lung tumor.
Drug: Pemetrexed 500 mg/m2 — Pemetrexed is an antifolate chemotherapeutic agent. In this study, it is specifically used for patients with non-squamous non-small cell lung cancer (NSCLC). It is administered intravenously at a dose of 500 mg/m² on Day 1 of each 3-week cycle. Patients receive 2 cycles of pemetrexed in combination with sintilimab (anti-PD-1 antibody) and carboplatin (platinum-based agent) as part of the neoadjuvant regimen. To reduce toxicity risks, standard premedication (including folic acid, vitamin B12 supplementation, and corticosteroids) is required as per the product label. This systemic chemotherapy phase is initiated within 7 days after the completion of stereotactic body radiotherapy (SBRT) to the primary lung tumor.
Radiation: Stereotactic body radiotherapy (SBRT) — Stereotactic Body Radiotherapy (SBRT) is a precise, high-dose form of external beam radiation therapy. In this study, SBRT is directed only at the primary lung tumor (not the lymph nodes). The treatment is delivered in 3 fractions (sessions) over approximately 3 days, with a total dose of 24 Gy (8 Gy per fraction). Treatment planning is based on 4D-CT simulation to account for respiratory motion. The SBRT is completed before the initiation of systemic therapy (sintilimab + chemotherapy).
Procedure: non-small cell lung cancer — Radical lung resection is the planned definitive treatment for eligible patients. Approximately 4 weeks after neoadjuvant therapy, patients first undergo cervical mediastinoscopy for contralateral lymph node assessment. Only those with negative pathology proceed to surgery 2 weeks later. The surgery involves initial video-assisted thoracoscopic dissection of remaining contralateral nodes (specific stations based on primary tumor side) with intraoperative frozen section. If negative, patients undergo immediate repositioning and radical lung resection (lobectomy/pneumonectomy) with ipsilateral lymphadenectomy(right side dissection of lymph nodes in groups 3A, 9R and 10R, left side dissection of lymph nodes in groups 5, 6, 9L and 10L).

SUMMARY:
This is a Phase II clinical trial evaluating the efficacy and safety of a new treatment approach for patients with locally advanced non-small cell lung cancer (NSCLC) that has spread to lymph nodes on the opposite side of the chest (known as N3 lymph node involvement).

The study will enroll 28 patients aged 18 to 75 years with previously untreated, potentially resectable NSCLC classified as stage IIIB-IIIC. Participants will receive a combination of stereotactic body radiation therapy (SBRT) to the primary lung tumor, followed by two cycles of sintilimab (an immunotherapy drug) plus platinum-based chemotherapy before surgery.

The main goals of the study are to see whether this treatment can shrink or eliminate cancer in the contralateral mediastinal lymph node (lymph node downstaging) and allow more patients to undergo curative surgery. Secondary goals include assessing pathological response rates, surgical outcomes, survival, and safety.

Patients will be closely monitored during and after treatment, with follow-up visits planned for up to 5 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary Participation: The patient volunteers to participate and signs a written informed consent form.
2. Pathology and Staging: Cytologically or histologically confirmed, previously untreated non-small cell lung cancer (NSCLC) with contralateral mediastinal lymph node involvement (N3), classified as stage IIIB or IIIC according to the 9th edition of the International Association for the Study of Lung Cancer (IASLC) staging manual. Baseline staging must be performed with either PET/CT or a combination of contrast-enhanced CT of chest/abdomen + bone scan + brain MRI.
3. Surgical Feasibility: The lung lesion is considered **potentially resectable as evaluated by a multidisciplinary team that includes a thoracic surgeon.
4. Performance Status: Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
5. Adequate Organ Function:

(1) Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L (2) Platelet count ≥ 100 x 10^9/L (3) Hemoglobin > 9.0 g/dL (4) Serum creatinine ≤ 1.5 x upper limit of normal (ULN) OR creatinine clearance (CrCl) ≥ 40 mL/min (5) Aspartate aminotransferase (AST)/Alanine aminotransferase (ALT) ≤ 3 x ULN (6) Total bilirubin ≤ 1.5 x ULN (7) Forced expiratory volume in 1 second (FEV1) ≥ 1.2 L or > 40% of predicted value (8) International normalized ratio (INR) and activated partial thromboplastin time (aPTT) within normal limits.

6. Age: Between 18 and 75 years old.

Exclusion Criteria

1. Autoimmune Disease: Active or suspected autoimmune disease. Exception: Patients with vitiligo, type I diabetes mellitus, or hypothyroidism requiring only hormone replacement therapy (e.g., Hashimoto's thyroiditis) with no signs of active disease may be enrolled.
2. Immunosuppressive Therapy: Requires systemic corticosteroid therapy (>10 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days prior to enrollment.
3. Prior Chest Radiotherapy: History of prior radiotherapy to the chest.
4. Active Bleeding: Presence of clinically significant active bleeding prior to treatment.
5. Severe Organ Dysfunction: Severe cardiac, pulmonary, hepatic, or renal dysfunction, hematopoietic system disease, or cachexia, as judged by the investigator to be intolerable to chemo-radiotherapy.
6. Poorly Controlled Diabetes: History of diabetes mellitus for >10 years with unsatisfactory glycemic control.
7. Interstitial Lung Disease: History of interstitial lung disease or non-infectious pneumonitis.
8. Driver Gene Mutations: NSCLC with known activating EGFR mutations or ALK fusion gene positivity.
9. Other Malignancies:

   Excluded: History of other active malignancies within the past 2 years, except for adequately treated non-melanoma skin cancer or carcinoma in situ (e.g., bladder, gastric, colorectal, endometrial, cervical, melanoma, or breast).

   Exception: Patients with other malignancies who have achieved complete remission for ≥2 years and do not require additional anti-tumor therapy during this study may be enrolled.
10. Compliance/Understanding: Medical, psychological, or physiological conditions that, in the investigator's judgment, prevent the patient from completing the study or understanding the study information.
11. Prior Immune Therapy: Previous treatment with any anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other drug targeting T-cell co-stimulation or checkpoint pathways.
12. Active Viral Infection:

(1) Active Hepatitis B (HBsAg positive AND HBV DNA ≥ 2000 IU/mL or 10^4 copies/mL).

(2) Active Hepatitis C (HCV antibody positive AND HCV RNA above the lower limit of detection).

13. HIV/AIDS: Known positive test for human immunodeficiency virus (HIV) or diagnosed acquired immunodeficiency syndrome (AIDS).

14. Allergy: Known history of hypersensitivity to sintilimab, any of the chemotherapy agents used, or any of their excipients.

15. Pregnancy/Lactation: Pregnant or breastfeeding women. 16. Metastatic Disease: Presence of supraclavicular lymph node metastasis or distant metastasis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2032-10-31 (Estimated)

PRIMARY OUTCOMES:
Contralateral Mediastinal Lymph Node Downstaging Rate | From the start of neoadjuvant therapy until post-surgical pathological assessment, approximately 12 weeks.
Surgical Conversion Rate | From the start of neoadjuvant therapy until post-surgical pathological assessment, approximately 12 weeks.

SECONDARY OUTCOMES:
Major Pathological Response Rate | At the time of surgical pathological assessment, approximately 12 weeks after the start of neoadjuvant therapy.
Pathological Complete Response Rate | At the time of surgical pathological assessment, approximately 12 weeks after the start of neoadjuvant therapy.
R0 Resection Rate | At the time of surgical pathological assessment, approximately 12 weeks after the start of neoadjuvant therapy.
Event-Free Survival | From enrollment until the first occurrence of an EFS event, assessed up to 5 years.
Overall Survival | From enrollment until death from any cause, assessed up to 5 years.
Incidence of Adverse Events | From the start of neoadjuvant therapy until 90 days after the last dose of study drug or 30 days after surgery, whichever is later.

IPD SHARING:
Plan to Share IPD: No